CLINICAL TRIAL: NCT01377571
Title: A Phase II, Randomized, Double-blind, Vaccine-controlled Dose-escalating Study to Evaluate the Immunogenicity, Reactogenicity and Safety of Oral Live Attenuated Human Rotavirus (HRV) Vaccine (Rotavin-M1) in Healthy Infants in Vietnam
Brief Title: A Dose-escalating Study to Evaluate the Immunogenicity and Safety of Rotavin-M1 Vaccine in Healthy Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Hygiene and Epidemiology, Vietnam (Other)
Collaborators: Center for Research and Production of Vaccines and Biologicals, Vietnam (Other Government)
Responsible Party: Principal Investigator, Dang Duc Anh, Director, National Institute of Hygiene and Epidemiology, Vietnam
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: Rotavin02; KC.10.33/06-10 (Other Grant/Funding Number: The Ministry of Science and Technology, Vietnam)
Record Dates: First submitted 2011-05-19; First posted 2011-06-21 (Estimated); Last update posted 2016-07-04 (Estimated); Status verified 2016-06

CONDITIONS: Diarrhea; Fever; Nausea; Vomit; Irritability
Keywords: diarrhea; fever; nausea; vomit; irritability
MeSH Terms: conditions — Diarrhea; Fever; Nausea; Vomiting | interventions — RIX4414 vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Rotavin2H (Experimental): 2 doses of Rotavin-M1 vaccine, 106.3FFU/dose, 2-month separation between doses
  Interventions: Biological: Rotarix
- Rotavin2L (Experimental): 2 doses of Rotavin-M1 vaccine, 106.0FFU/dose, 2-month interval between doses
  Interventions: Biological: Rotarix
- Rotavin3H (Experimental): 3 doses of Rotavin-M1 vaccine, 106.3FFU/dose, 1-month interval between doses
  Interventions: Biological: Rotarix
- Rotavin3L (Experimental): 3 doses of Rotavin-M1, 106.0FFU/dose, 1-month interval between doses
  Interventions: Biological: Rotarix

INTERVENTIONS:
Biological: Rotarix — 2 doses of Rotarix vaccine, 106.5CID/dose, 1-month interval between doses
  Other Names: RotarixTM, GSK biologicals

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of Rotavin-M1 produced by the Center for Research and Production of Vaccines and Biologicals (POLYVAC) in infants in Vietnam. In addition, we evaluate different dosages and schedules to determine the best regimen to test in a clinical trial.

DETAILED DESCRIPTION:
Rotavirus (RV) is the most important cause of acute gastroenteritis in children worldwide. In Vietnam rotavirus causes an estimated 122,000-140,000 hospitalizations and 2900-5400 deaths per year among children under 5 years of age (1). Over the past 13 years, sentinel hospital surveillance identified rotavirus in 44%-62% of children admitted for the treatment of acute diarrhea in Vietnam (2-4). Such a high burden of disease justified accelerated development of a new and locally manufactured vaccine against rotavirus in Vietnam. It is estimated that if a vaccine was introduced in the current childhood immunization schedule, it could reduce severe rotavirus disease by about 60% or more given current vaccine efficacies and coverage (5).

The Government of Vietnam has pursued a policy to encourage local vaccine production so the country could be self-reliant with affordable vaccines for its population (6). Over the past decades, several locally produced vaccines for poliomyelitis, cholera, Japanese encephalitis, and Diphtheria-Pertussis-Tetanus have contributed to the reduction in the prevalence of these diseases and to the eradication of polio over the past decade. While two commercial rotavirus vaccines, RotarixTM (GSK, Belgium) and RotaTeq® (Merck), have both been tested in Vietnam, neither is currently available at an affordable cost for the national program. Therefore, the candidate vaccine, Rotavin-M1, was developed in order to fill this need for a more affordable vaccine for Vietnamese children (6). This vaccine is similar to RotarixTM, and was developed by selecting a common G1P[8] strain and attenuating it through serial passages and plaque purification in qualified Vero cells under GLP conditions.

ELIGIBILITY:
Inclusion Criteria:

* At dose 1

  1. A healthy male or female, 6 to 12 weeks of age (42 days to 84 days of age).
  2. Full term gestation (>=37 weeks).
  3. Birth weight of the subject should be >=2.5 kg.
  4. Healthy subjects as established by medical history and clinical examination before entering into the study.
  5. Did not use any dose of Rota virus vaccine.
  6. Written informed consent obtained from the parent or guardian of the subject.
* At dose 2

  1. Received dose 1.
  2. Oral informed consent obtained from the parent or guardian of the subject for continuing participate the study.
* At dose 3

  1. Received both dose 1 and dose 2.
  2. Oral informed consent obtained from the parent or guardian of the subject for continuing participate the study.

Exclusion Criteria:

* At dose 1

  1. Has a chronic disease (cardiovascular, liver, kidney disease).
  2. Acute disease at the time of enrolment.
  3. Administering corticosteroids (> 1mg/kg/day).
  4. Received any immunosuppressive therapy within 4 week before vaccination (Administration of immunoglobulins and/or any blood product or corticosteroids for >2 weeks).
  5. Immunosuppressive or immunodeficient condition.
  6. Family has immunosuppressive or immunodeficient condition medical history.
  7. History of high fever convulsion.
  8. Allergic or reaction with any component of vaccine, includes anaphylactic shock with any antibiotic.
  9. Preterm of gestation delivery (gestation period < 37 weeks).
  10. Low birth weight (<2.5 kg).
  11. Fever (axillary temperature >38oC) within 3 days before or on the day of vaccination.
  12. Malnutrition.
  13. Has any type of blood disorder, leukemia, or malignant tumor which can affect the bone marrow or lymph system.
  14. Use of any investigational or non-registered product (unlicensed drug or vaccine) other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* At dose 2

  1. Acute disease at the time of 2nd dose.
  2. Administering corticosteroids (> 1mg/kg/day).
  3. Received any immunosuppressive therapy within 4 week before vaccination (Administration of immunoglobulins and/or any blood product or corticosteroids for >2 weeks).
  4. History of allergic disease or reactions likely to be exacerbated by any component of the study vaccine.
  5. Fever (axillary temperature >38oC) within 3 days before or on the day of vaccination.
  6. Has any type of blood disorder, leukemia, or malignant tumor which can affect the bone marrow or lymph system.
  7. Use of any investigational or non-registered product (unlicensed drug or vaccine) other than the study vaccine during the study period.
* At dose 3

  1. Acute disease at the time of 3rd dose.
  2. Administering corticosteroids (> 1mg/kg/day).
  3. Received any immunosuppressive therapy within 4 week before vaccination (Administration of immunoglobulins and/or any blood product or corticosteroids for >2 weeks).
  4. History of allergic disease or reactions likely to be exacerbated by any component of the study vaccine.
  5. Fever (axillary temperature >38oC) within 3 days before or on the day of vaccination.
  6. Has any type of blood disorder, leukemia, or malignant tumor which can affect the bone marrow or lymph system.
  7. Use of any investigational or non-registered product (unlicensed drug or vaccine) other than the study vaccine during the study period.

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2009-10; Primary Completion 2010-03 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
To assess immunogenicity of a new rotavirus vaccine Rotavin-M1 in terms of anti-rotavirus IgA antibody seroconversion 1 month after complete the vaccination schedule | up to 7 months
  To assess immunogenicity of Rotavin-M1 of 2 titers (10e6.0 and 10e6.3FFU/dose) and 2 schedules (3 doses and 1-month interval between vs 2 doses and 2-month interval between doses), compared with 2 doses GSK's lyophilized Rotarix (10e6.5 CID50/dose).

SECONDARY OUTCOMES:
To assess immunogenicity of Rotavin-M1 vaccine versus GSK Biologicals' HRV vaccine in terms of anti-rotavirus IgA antibody seroconversion at Month 2 in the group receiving the vaccines. | up to 7 months
  To assess immunogenicity of Rotavin-M1 vaccine (of different dosages and schedules) versus GSK Biologicals' HRV vaccine in terms of anti-rotavirus IgA antibody seroconversion at Month 2 in the group receiving the vaccines.
To assess immunogenicity of Rotavin-M1 vaccine versus GSK Biologicals' HRV vaccine in terms of anti-rotavirus IgA antibody GMT at Month 2 in the group receiving the vaccines. | up to 7 months
  To assess immunogenicity of Rotavin-M1 vaccine (of different dosages and schedules) versus GSK Biologicals' HRV vaccine in terms of anti-rotavirus IgA antibody GMT at Month 2 in the group receiving the vaccines.
To assess immunogenicity of Rotavin-M1 vaccine versus GSK Biologicals' HRV vaccine in terms of anti-rotavirus IgA antibody GMT at Month 3 in the group receiving the vaccines. | up to 7 months
  To assess immunogenicity of Rotavin-M1 vaccine (of different dosages and schedules) versus GSK Biologicals' HRV vaccine in terms of anti-rotavirus IgA antibody GMT at Month 3 in the group receiving the vaccines.
To assess the safety and reactogenicity of each dose of Rotavin-M1 versus GSK's biologicals Rotarix | up to 7 months
  To assess immediate reactions (30minutes) after administration of each dose To assess adverse events 30 days after each dose To assess change in blood cell counts (red blood cells, white blood cells, platelets), blood urea nitrogen concentration, transaminase concentration (ALT, AST)
To assess the presence of rotavirus (RV) in GE stools collected after administration of first dose of the study vaccine up to 1 month after the last dose. | up to 7 months
  To assess the presence of rotavirus (RV) in GE stools collected after administration of the first dose of the study vaccine up to 1 month after the last dose.
To assess the shedding of rotavirus (RV) in stools collected daily for 7 days after administration of each dose of the study vaccine. | up to 7 months
  To assess the shedding of rotavirus (RV) in stools collected daily for 7 days after administration of each dose of the study vaccine
To compare the RV antibody titers 1 year after the first doses between one Rotavin-M1 group and Rotarix | up to 15 months
  To assess the RV antibody titers 1 year after the 1st dose between Rotavin-M1 group (106.3FFU/dose, 2 doses, 2-month interval) and Rotarix group (106.0CID/dose, 2 doses, 1-month interval between doses).

CONTACTS AND LOCATIONS:
Overall Officials: Anh D Dang, PhD., Principal Investigator — The National Institute of Hygiene and Epidemiology; Thiem D Vu, MD., PhD., Principal Investigator — The National Institute of Hygiene and Epidemiology
Locations (1):
- Preventive Medicine center, Thanh Sơn, Phu Tho, Vietnam

REFERENCES:
- [Background] Anh DD, Thiem VD, Fischer TK, Canh DG, Minh TT, Tho le H, Van Man N, Luan le T, Kilgore P, von Seidlein L, Glass RI. The burden of rotavirus diarrhea in Khanh Hoa Province, Vietnam: baseline assessment for a rotavirus vaccine trial. Pediatr Infect Dis J. 2006 Jan;25(1):37-40. doi: 10.1097/01.inf.0000195635.05186.52. PMID 16395100
- [Background] Van Man N, Luan le T, Trach DD, Thanh NT, Van Tu P, Long NT, Anh DD, Fischer TK, Ivanoff B, Gentsch JR, Glass RI; Vietnam Rotavirus Surveillance Network. Epidemiological profile and burden of rotavirus diarrhea in Vietnam: 5 years of sentinel hospital surveillance, 1998-2003. J Infect Dis. 2005 Sep 1;192 Suppl 1:S127-32. doi: 10.1086/431501. PMID 16088796
- [Background] Ngo TC, Nguyen BM, Dang DA, Nguyen HT, Nguyen TT, Tran VN, Vu TT, Ogino M, Alam MM, Nakagomi T, Nakagomi O, Yamashiro T. Molecular epidemiology of rotavirus diarrhoea among children in Haiphong, Vietnam: the emergence of G3 rotavirus. Vaccine. 2009 Nov 20;27 Suppl 5:F75-80. doi: 10.1016/j.vaccine.2009.08.074. PMID 19931725
- [Background] Nguyen TA, Yagyu F, Okame M, Phan TG, Trinh QD, Yan H, Hoang KT, Cao AT, Le Hoang P, Okitsu S, Ushijima H. Diversity of viruses associated with acute gastroenteritis in children hospitalized with diarrhea in Ho Chi Minh City, Vietnam. J Med Virol. 2007 May;79(5):582-90. doi: 10.1002/jmv.20857. PMID 17385670
- [Background] Kim SY, Goldie SJ, Salomon JA. Cost-effectiveness of Rotavirus vaccination in Vietnam. BMC Public Health. 2009 Jan 21;9:29. doi: 10.1186/1471-2458-9-29. PMID 19159483
- [Background] Luan le T, Trang NV, Phuong NM, Nguyen HT, Ngo HT, Nguyen HT, Tran HB, Dang HN, Dang AD, Gentsch JR, Wang Y, Esona MD, Glass RI, Steele AD, Kilgore PE, Nguyen MV, Jiang B, Nguyen HD. Development and characterization of candidate rotavirus vaccine strains derived from children with diarrhoea in Vietnam. Vaccine. 2009 Nov 20;27 Suppl 5:F130-8. doi: 10.1016/j.vaccine.2009.08.086. PMID 19931712
- [Derived] Dang DA, Nguyen VT, Vu DT, Nguyen TH, Nguyen DM, Yuhuan W, Baoming J, Nguyen DH, Le TL; Rotavin-M1 Vaccine Trial Group. A dose-escalation safety and immunogenicity study of a new live attenuated human rotavirus vaccine (Rotavin-M1) in Vietnamese children. Vaccine. 2012 Apr 27;30 Suppl 1:A114-21. doi: 10.1016/j.vaccine.2011.07.118. PMID 22520120